CLINICAL TRIAL: NCT03585660
Title: MRI Derived Quantitative Risk Maps for Prostate Cancer Diagnosis Using Targeted Biopsy
Brief Title: Developing an Imaging-Based Tool to Identify Areas for Prostate Cancer Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB17-1694
Record Dates: First submitted 2018-06-19; First posted 2018-07-13 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Interventional Arm (Experimental): Participants will undergo diagnostic MRI exam followed by clinical biopsies of suspected prostate cancer tumors.
  Interventions: Procedure: Diagnostic MRI; Procedure: Diagnostic Prostate Biopsy; Device: Risk Map DSS tool

INTERVENTIONS:
Procedure: Diagnostic MRI — Participants will be scanned using a standard clinical prostate MRI protocol.
Procedure: Diagnostic Prostate Biopsy — Participants will undergo a prostate biopsy as their standard of care treatment. The provider performing biopsy will select areas to be biopsies as part of normal clinical judgment.
Device: Risk Map DSS tool — The Risk Map DSS tool will select up to 2 additional areas to be biopsied based on analysis of MRI images. The clinical provider will make final decision on areas to be biopsied.

SUMMARY:
The purpose of the proposed research is to test and validate a Risk Map decision-support system (DSS) for prostate cancer Magnetic Resonance Imaging (MRI) interpretation and identification of clinically significant tumor site(s).

ELIGIBILITY:
Inclusion Criteria:

* Patients with known or suspected prostate cancer who have been referred to the Department of Radiology at the University of Chicago Medical Center for a diagnostic MRI exam of the prostate, to be followed by an MRI-guided fusion biopsy of the prostate.
* Written informed consent.

Exclusion Criteria:

* Patients incapable of giving informed written consent;
* Patients who cannot adhere to the experimental protocols for any reason, or have an inability to communicate with the researcher;
* Patients with psychiatric disorders that affect their ability to consent for themselves will be excluded and not the entire population of patients with psychiatric disorders.
* Prisoners;
* Minor children (under the age of 18 years old).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aytekin Oto, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chatterjee A, Yousuf AN, Engelmann R, Harmath C, Lee G, Medved M, Jamison EB, Lorente Campos A, Gundogdu B, Gerber G, Reynolds LF, Modi PK, Antic T, Giurcanu M, Eggener S, Karczmar GS, Oto A. Prospective Validation of an Automated Hybrid Multidimensional MRI Tool for Prostate Cancer Detection Using Targeted Biopsy: Comparison with PI-RADS-based Assessment. Radiol Imaging Cancer. 2025 Jan;7(1):e240156. doi: 10.1148/rycan.240156. PMID 39836080

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 106 patients were enrolled in the study. Patients were recruited based on physician referral at UChicago Medical Center. The 1st patient was enrolled on August 28, 2018, and the last patient was enrolled on March 29, 2023.
Pre-assignment Details: 112 patients were screened and 6 patients did not meet eligibility criteria of the study.
Period: Overall Study
Arm/Group | Interventional Arm
Started | 106
Completed | 91
Not Completed | 15
Not completed — operator error | 1
Not completed — technical error | 2
Not completed — hip prosthesis | 2
Not completed — did not undergo biopsy | 8
Not completed — scanner problem | 2

BASELINE CHARACTERISTICS:
Arm/Group | Interventional Arm
Number analyzed (Participants) | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.44 (7.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 106
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4
  Black | 27
  Hispanic | 8
  Unknown | 4
  White | 63
Prostate Specific Antigen (PSA) [Mean (Standard Deviation); unit: ng/mL] | 8.81 (11.69)

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of HM-MRI
Description: The accuracy of HM-MRI is defined as the proportion of correctly diagnosed participants for prostate cancer using HM-MRI.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Interventional Arm
Number analyzed (Participants) | 91
proportion of participants | 0.55 [0.45 to 0.65]
Statistical Analysis 1: Comparison: Interventional Arm; The null hypothesis is that the accuracy of HM-MRI and mp-MRI are the same and the alternative hypothesis is that the accuracy of HM-MRI is greater than the accuracy of mp-MRI; Test type: Superiority; p = 0.02, bootstrap z-test; The standard error of the difference in accuracy was estimated using nonparametric bootstrap, with B=9999 resamples

2. Primary Outcome: Area Under the ROC Curve (AUC) of HM-MRI
Description: In the case of a binary predictor (HM-MRI), the area under a receiver operating characteristic (ROC) curve is equivalent to the average of sensitivity and specificity. The area under an ROC curve ranges from 0 to 1.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: probability
Arm/Group | Interventional Arm
Number analyzed (Participants) | 91
probability | 0.63 [0.52 to 0.74]
Statistical Analysis 1: Comparison: Interventional Arm; The null hypothesis is that the AUCs of HM-MRI and mp-MRI are the same and the alternative hypothesis is that the AUC of HM-MRI is greater than the AUC of mp-MRI; Test type: Superiority; p = 0.08, bootstrap z-test; The standard error of the difference of AUCs was estimated using nonparametric bootstrap, with B=9999 resamples

3. Secondary Outcome: Sensitivity of HM-MRI
Description: Sensitivity of HM-MRI is defined as the proportion of participants who were found positive of prostate cancer using HM-MRI among the participants who were found positive of prostate cancer using biopsy.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Interventional Arm
Number analyzed (Participants) | 91
proportion of participants | 0.91 [0.81 to 1]
Statistical Analysis 1: Comparison: Interventional Arm; The null hypothesis is that the sensitivity of HM-MRI and mp-MRI are the same and the alternative hypothesis is that the sensitivity of HM-MRI is greater than the sensitivity of mp-MRI; Test type: Superiority; p = 0.97, bootstrap z-test

4. Secondary Outcome: Specificity of HM-MRI
Description: Specificity of HM-MRI is defined as the proportion of participants who were found negative of prostate cancer using HM-MRI among the participants who were found negative using biopsy.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Interventional Arm
Number analyzed (Participants) | 91
proportion of participants | 0.36 [0.23 to 0.48]
Statistical Analysis 1: Comparison: Interventional Arm; The null hypothesis is that the specificity of HM-MRI and mp-MRI are the same and the alternative hypothesis is that the specificity of HM-MRI is greater than the specificity of mp-MRI; Test type: Superiority; p < 0.01, bootstrap z-test

5. Secondary Outcome: Positive Predictive Value (PPV) of HM-MRI
Description: Positive predictive value (PPV) of HM-MRI is defined as the proportion of participants who were found positive of prostate cancer using biopsy among the participants who were found positive using HM-MRI.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Interventional Arm
Number analyzed (Participants) | 91
proportion of participants | 0.43 [0.31 to 0.55]
Statistical Analysis 1: Comparison: Interventional Arm; Test type: Superiority — The null hypothesis is that the PPV of HM-MRI and mp-MRI are the same and the alternative hypothesis is that the PPV of HM-MRI is greater than the PPV of mp-MRI; p = 0.06, bootstrap z-test

6. Secondary Outcome: Negative Predictive Value (NPV) of HM-MRI
Description: Negative predictive value (NPV) of HM-MRI is defined as the proportion of participants who were found negative of prostate cancer using biopsy among the participants who were found negative using HM-MRI.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Interventional Arm
Number analyzed (Participants) | 91
proportion of participants | 0.88 [0.74 to 1]
Statistical Analysis 1: Comparison: Interventional Arm; Test type: Superiority — The null hypothesis is that the NPV of HM-MRI and mp-MRI are the same and the alternative hypothesis is that the NPV of HM-MRI is greater than the NPV of mp-MRI; p = 0.97, bootstrap z-test

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Interventional Arm
All-Cause Mortality (participants affected / at risk) | 0/106
Serious Adverse Events (participants affected / at risk) | 0/106
Other Adverse Events (participants affected / at risk) | 0/106

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/60/NCT03585660/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-28): https://cdn.clinicaltrials.gov/large-docs/60/NCT03585660/ICF_001.pdf